CLINICAL TRIAL: NCT05927818
Title: Efficacy of Sentinel Lymph Node Biopsy in Early-Stage Ovarian Cancer
Brief Title: Sentinel Lymph Node Biopsy in Early-Stage Ovarian Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mustafa Albayrak, MD, Gynecologic Oncology Fellow, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1740514
Record Dates: First submitted 2023-06-09; First posted 2023-07-03 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Sentinel Lymph Node; Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Intervention Model Description: A single arm interventional study aiming at the detection of the effectiveness of sentinel lymph node biopsy compared to systemic lymphadenectomy in participants who has high suspicion of an adnexal mass for early ovarian cancer clinically before operation in a single center. Clinical exam, radiological evaluation and tumor markers are primary determinants in using an adnexal mass to be assigned as 'highly suspicious'. The interventional and control arms are the same participant (each participant becomes its own control since the sentinel node biopsy- interventional arm - results are to be compared to systematic lymphadenectomy -control arm- results). Intervention is injection of 2-4 mL sterile charcoal to the infundibulopelvic ligament or mesovarium of the suspicious adnexal mass followed by collection of stained sentinel lymph nodes and lymph nodes by systematic lymphadenectomy.
Masking Description: No party in our clinical trial are prevented from having knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sentinel Lymph Node Biopsy and Systematic Lymph Node Dissection (Single Arm) (Experimental): This is a single arm interventional study in which the interventional and control arms are the same participant (each participant becomes its own control since the sentinel node biopsy- interventional arm - results are to be compared to systematic lymphadenectomy results-control arm). Intervention is injection of 2-4 mL sterile charcoal to the infundibulopelvic ligament or mesovarium of the suspicious adnexal mass followed by collection of stained sentinel lymph nodes and lymph nodes by systematic lymphadenectomy.
  Interventions: Diagnostic Test: Sentinel lymph node biopsy (using sterile charcoal stain) in early ovarian cancer

INTERVENTIONS:
Diagnostic Test: Sentinel lymph node biopsy (using sterile charcoal stain) in early ovarian cancer — Described in previous sections
  Other Names: Systematic lymphadenectomy

SUMMARY:
The primary goal of this prospective study is to define the efficacy of the sentinel lymph node biopsy (SLNB) procedure by comparing it to the results obtained from systematic lymphadenectomy, each performed in participants with a suspicious adnexal mass for early-stage ovarian cancer.

DETAILED DESCRIPTION:
Ovarian cancer is the leading cause of mortality among gynecologic cancers. Although most women are diagnosed at advanced stage, about 20% are can be diagnosed at an earlier stage. Treatment and prognosis depends on the correct assessment of stage of the apparently early stage (Stage I and II). About 10-30% of apparently early stage ovarian cancer patients are upstaged based on the final pathology report. Detection of positive lymph node is an important contributor for upstaging of apparently early stage ovarian cancer. However, systematic lymphadenectomy carries immediate and long term risks for patients including bleeding, massive transfusions, prolongation of operation time, serious major vessel and major abdominal organ injury and death. These risks are especially increased in paraaortic lymphadenectomy which is an integral part of staging procedure in early ovarian cancer.

Sentinel lymph node biopsy (SLNB) procedure is the biopsy of one or two lymph node(s) which represents the lymph node basin draining the area of malignancy. This biopsy may potentially eliminate the need systemic pelvic / paraaortic lymphadenectomy. Although SLNB became an integral and accepted procedure in endometrium and cervix cancers, available data on the SLNB for ovarian cancer is limited and is in its infancy to be incorporated in routine practice of ovarian cancer surgery.

So, investigators aim to compare the effectiveness of SLNB procedure results with systematic lymphadenectomy, both performed in each participant, either by laparotomy or laparoscopy.

Technically, 2-4 mL of sterile black carbon stain is carefully injected beneath the adnexal mass just under peritoneal covering of mesovarium or infundibulopelvic ligament avoiding intravascular injection before removal of suspicious adnexal mass for frozen section. This is done classically through a laparotomy incision but can also be performed laparoscopically via a needle introduced transcutaneously into the base of adnexa under optical supervision. 10-15 minute interval is allowed before resection of adnexal mass for frozen section. A peritoneal incision and pelvic and paraaortic retroperitoneal dissection is carried out for identification of major vessels and important surgical landmarks (abdominal ureters, gonadal vessels, inferior mesenteric artery and etc.) up to the left renal vein to visually detect the sentinel lymph node(s) stained in black. Lymphatic vessels are carefully eliminated visually not to be biopsied instead of sentinel lymph node. An additional 2 mL injection is allowed if a SLN could not be detected before systematic lymphadenectomy, adnexectomy and other surgical staging procedures. Frozen section of a adnexal mass is carried out thereafter following the detection and biopsy of SLN. Systematic lymphadenectomy is abandoned in case of a non-malignant frozen section result.

ELIGIBILITY:
Inclusion Criteria:

Must have a suspicious adnexal mass for early stage ovarian cancer

Must be medically and surgically fit enough to perform SLNB and complete the systematic lymphadenectomy.

-

Exclusion Criteria:

Ovarian mass with low probability for early stage ovarian cancer.

Medical or surgical contraindications for surgical comprehensive staging.

Metastatic cancers or double primary cancers (metachronous) of ovary

Recurrent ovarian cancer

Preoperative or intraoperative finding of advanced ovarian cancer (FİGO stage III and IV)

Neoadjuvant ovarian cancer

-

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy of sentinel lymph node biopsy in highly suspicious adnexal masses for early-stage ovarian cancer | From the day of surgery to final pathology report (two weeks)
  Sensitivity, specificity, positive and negative predictive value for sentinel lymph biopsy results (compared to lymph nodes collected by systemic lenfadenopathy) will be calculated. These calculations will be expressed in percentages and will be compared using appropriate statistical method.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey, Turkey (Türkiye)

REFERENCES:
- [Background] Negishi H, Takeda M, Fujimoto T, Todo Y, Ebina Y, Watari H, Yamamoto R, Minakami H, Sakuragi N. Lymphatic mapping and sentinel node identification as related to the primary sites of lymph node metastasis in early stage ovarian cancer. Gynecol Oncol. 2004 Jul;94(1):161-6. doi: 10.1016/j.ygyno.2004.04.023. PMID 15262135
- [Background] Hassanzadeh M, Hosseini Farahabadi E, Yousefi Z, Kadkhodayan S, Zarifmahmoudi L, Sadeghi R. Lymphatic mapping and sentinel node biopsy in ovarian tumors: a study using intra-operative Tc-99m-Phytate and lymphoscintigraphy imaging. J Ovarian Res. 2016 Sep 7;9(1):55. doi: 10.1186/s13048-016-0265-4. PMID 27604260
- [Background] Uccella S, Nero C, Vizza E, Vargiu V, Corrado G, Bizzarri N, Ghezzi F, Cosentino F, Turco LC, Fagotti A, Scambia G. Sentinel-node biopsy in early-stage ovarian cancer: preliminary results of a prospective multicentre study (SELLY). Am J Obstet Gynecol. 2019 Oct;221(4):324.e1-324.e10. doi: 10.1016/j.ajog.2019.05.005. Epub 2019 May 10. PMID 31082385
- [Background] Lago V, Bello P, Montero B, Matute L, Padilla-Iserte P, Lopez S, Marina T, Agudelo M, Domingo S. Sentinel lymph node technique in early-stage ovarian cancer (SENTOV): a phase II clinical trial. Int J Gynecol Cancer. 2020 Sep;30(9):1390-1396. doi: 10.1136/ijgc-2020-001289. Epub 2020 May 23. PMID 32448808
- [Background] Vanneuville G, Mestas D, Le Bouedec G, Veyre A, Dauplat J, Escande G, Guillot M. The lymphatic drainage of the human ovary in vivo investigated by isotopic lymphography before and after the menopause. Surg Radiol Anat. 1991;13(3):221-6. doi: 10.1007/BF01627990. PMID 1754957